CLINICAL TRIAL: NCT02340377
Title: Core Body Temperature During Hyperthermia in a Whole Body Hyperthermia Device (Heckel HT 3000): Monitoring Core Body Temperature Using Wireless Technology
Brief Title: Pill Study Hyperthermia Device (Heckel HT 3000): Monitoring Core Body Temperature Using Wireless Technology
Status: Terminated | Type: Observational
Why Stopped: investigator transferred institutions
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Charles (Chuck) Raison, Professor, Department of Psychiatry; College of Medicine, University of Arizona
Other Study IDs: 14-11566-046
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Core Body Temperature
Keywords: core body temperature; whole-body hyperthermia; rectal body temperature

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ELITE 3 HQ — The pill is about the size of a multivitamin, is coated with special medical plastic, and is easy to swallow. The pill sends radio signals to a small recording device that participants wear that send a signal to a monitor and records the participant's internal body temperature. The pill will exit the participant's body in one of his/her bowel movements approximately 1-5 days after ingestion. Pills are not reused.
  Other Names: Core body temperature indigestible measuring device

SUMMARY:
The primary objective of the proposed study is to determine the use of a wireless method to monitor and record core body temperature during a Whole Body Hyperthermia treatment, compared to an indwelling rectal thermometer.

This protocol is intended to study the differences between a rectal temperature probe and an approved wireless and indigestible thermometer during a WBH session. The current standard in monitoring core body temperature is the usage of an indwelling rectal thermometer. Many patients and potential study subjects, however, decline receiving the treatment, due to the discomfort of using this measuring method and a wireless measuring device would open the possibility for those patients to receive a treatment. The primary endpoint for example of a treatment for MDD is currently defined with reaching a rectal temperature of 38.5 C. However, due to the proximity of the probe to the body's surface, the core body temperature will vary from the rectal temperature and the comparison between the two methods with a validation of the wireless device is necessary.

The investigators will monitor subject's physiological outcome from a single Whole Body Hyperthermia treatment in an open fashion (no placebo/control condition). This study will include safety assessments 7 days several days prior to or same day as the WBH, and include follow-up assessments 1 day and 1 week later.

DETAILED DESCRIPTION:
This protocol will allow for the evaluation of a wireless measuring device for core body temperature and a comparison to the data taken with a rectal thermometer, during a Whole Body Hyperthermia (WBH) in various subject populations. The primary objective of the proposed study is a potential change from wired core body temperature measurement with a rectal thermometer to an indigestible thermometer with wireless technology.

The recent standard for measuring core body temperature during WBH procedures is the use of an indwelling rectal thermometer to constantly monitor the temperature for safety and for research reasons. Experiences from different clinics and research groups, including ours, show a high drop-out rate of potential study participants and patients, because of the discomfort of self-inserting a rectal thermometer for the treatment in a Whole-Body Hyperthermia. A wireless and reliable measuring technology would open this treatment for participants, who are declining their participation due to the indwelling thermometer. This device will exit the subject's body via bowel movement 1-5 days following ingestion and will not be reused.

Due to the proximity of the indwelling thermometer to the surface of the body, the temperature does not reflect the real core body temperature and preliminary data, taking by our group, suggest a significant, but stable difference between core body temperatures measured with an indigestible device, compared to the temperature taken with the rectal probe. WBH treatments, currently studied by our group at the University of Arizona, are of mild nature and the constant infra-red heating is stopped, as soon as a patient reaches the rectal temperature of 38.5 C. Due to the fact, that the bodies surface is heated up through the infrared exposure, the investigators assume, that the core body temperature will be lower, compared to the rectal temperature. A validation study in 20 subjects therefore is necessary to determine the differences in the measuring methods. This is especially important, as the end-point of the treatments is defined by the core body temperature, and different endpoints by switching from one measuring method to the other, without validation, would potentially bias the study results.

Receiving a treatment in the WBH machine is of non-significant risk and can be compared to e.g. a sauna visit or an intense exercise, in terms of the physiological reaction. It is currently studied by our group for the treatment of Major Depressive Disorder, PTSD and other chronic illnesses. This trial however will not be limited to only include individuals with MDD or PTSD, but will allow for an expanded use in all populations (while still excluding subjects based on safety parameters). The investigators will monitor subject's physiological and clinical outcomes (if applicable) from a single Whole Body Hyperthermia treatment in an open fashion (no placebo/control condition). This study will include safety assessments several days prior to or same day as the WBH, and include follow-up assessments 1 day and 1 week later.

ELIGIBILITY:
Inclusion Criteria:

* Male or females aged 18-50 years.
* Able to understand the nature of the study and able to provide written informed consent prior to conduct of any study procedures.
* Able to communicate in English with study personnel.
* For women of child-bearing potential (i.e., one who is biologically capable of become pregnant,) must be willing to use a medically acceptable form of birth control or practice abstinence for the duration of her participation in the trial per self-report.

Exclusion Criteria:

* Any of the following diagnoses, as identified by the psychiatric evaluation or study assessments:
* A current DSM-IV-TR Axis I diagnosis of Dementia; or
* Any current DSM-IV-TR Axis II diagnosis (i.e. personality disorder) that would suggest potential noncompliance with the protocol; or
* A lifetime history of Schizophrenia, Schizoaffective Disorder, or a Bipolar Disorder Type 1; or
* A diagnosis claustrophobia severe enough that it would impair ability to be in the Heckel HT3000 hyperthermia device
* A current (or within 6 months prior to the Screening visit) diagnosis of Anorexia Nervosa or Bulimia Nervosa
* Individuals with psychiatric diagnoses may be excluded per the investigator's discretion.
* If patient has a medical condition or disorder that:
* Is unstable and clinically significant, or:
* Could, in the investigator's opinion, interfere with the accurate assessment of safety or efficacy of the procedure, including:

  1. individuals who are using prescription drugs that may impair thermoregulatory cooling,
  2. individuals with cardiovascular conditions or problems (uncontrolled hypertension, congestive heart failure, or documented evidence of coronary artery disease)
  3. individuals with chronic conditions/diseases associated with a reduced ability initiate thermoregulatory cooling, including Parkinson's, multiple sclerosis, central nervous system tumors, and diabetes with neuropathy,
  4. individuals with a fever the day of study intervention (if so, they will be rescheduled),
  5. individuals with hypersensitivity to heat,
  6. individuals with enclosed infections, be they dental, in joints, or in any other tissues,
* Use of any psychotropic medications for 2 weeks (8 weeks for fluoxetine) prior to initiation of the study, with the exception of a stable dosage of benzodiazepine or non-benzodiazepine hypnotic medications (e.g. zolpidem (Ambien), zaleplon (Sonata), eszopiclone (Lunesta), lorazepam (Ativan), diazepam (Valium), clonazepam (Klonopin), alprazolam (Xanax),
* Women who are pregnant (HCG pregnancy test at screening, or lactating, or who plan to become pregnant during the study.
* Reasonable likelihood for non-compliance with the protocol for any other reason, in the opinion of the Investigator, prohibits enrollment of subject into the study.
* Obesity and overall size of subject. It will be up to the PI's discretion will consider BMI, waist circumference, and body fat composition when determining eligibility and safety of the individual.
* History of peripheral circulatory disease, for example peripheral vascular disease, deep vein thrombosis (DVT), or lymphedema.
* History of a cerebral vascular accident
* History of stroke, epilepsy or cerebral aneurisms
* Cancer in the last five years, except for fully resected non-melanoma skin cancer.
* Diabetes mellitus types I or II.
* Any clinically significant autoimmune disease (compensated hypothyroidism and fibromyalgia allowed)
* Active alcohol/drug abuse in 2 weeks prior to screening for those who have been dependent or have abused on drugs/alcohol in the last 2 months (with the exception of marijuana use).
* Individuals with a history of having difficulty swallowing food or large capsules will be excluded from participating in the assessment of core body temperature (because swallowing a large sensor pill is required). The indigestible temperature capsules will not be used in subjects with any known or suspected obstructive disease of the gastrointestinal tract including, but not limited to esophageal stricture, diverticulosis and inflammatory bowel disease (IBD), peptic ulcer disease, Crohn's disease, ulcerative colitis; previous gastrointestinal surgery.
* Individuals who have experience with cognitive enhancing programs such as Luminosity, Cogmed or Elevate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For the purposes of this study we will enroll subjects 18-50 years of age to undergo a Hyperthermia session in an open fashion. We expect approximately 20 - 30 subjects to undergo this open hyperthermia treatment. Subjects must be medically healthy enough to be able to undergo the Hyperthermia session, all exclusion criteria listed below address what is deemed "medically healthy", per self-report by potential subjects. There will be no inclusion of children, pregnant women, mentally impaired individuals, or prisoners in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Difference in core body temperature | WBH Heating Session (this takes place at the hospital and lasts approximately 2.5 hours)
  Core body temperature differences as measured by 1) a rectal temperature probe and 2) an approved wireless and indigestible thermometer during a WBH session.

SECONDARY OUTCOMES:
Change in Score on the Q-LESQ-SF (Quality of Life Enjoyment and Satisfaction Questionnaire -Short form) | WBH treatment day and 1 day following WBH treatment
  Percent change in scores between baseline and subsequent assessments will be assessed to determine the effect of WBH on self-reported quality of life.
Change in Score on the Positive and Negative Association Scale (PANAS) | During the WBH Session
  Percent change in scores on the PANAS Scale to assess the transient and fluctuating active mood states during the WBH procedure.
Change in Score on Cognition Tests | WBH treatment day and 1 day following WBH treatment

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Arizona, Department of Psychiatry, College of Medicine; Clemens Janssen, MS, Study Director — University of Arizona, Department of Psychiatry, College of Medicine
Locations (1):
- University of Arizona, Tucson, Arizona, United States